CLINICAL TRIAL: NCT03684954
Title: Prf Controlled, Randamized Clinical Trial of THE EFFECT OF PLATELET RICH FIBRIN( PRF ) VERSUS XENOGRAFT IN CLOSED SINUS LIFT AND IMLANT PLACEMENT ON IMPLANT STABILITY IN PATIENTS WITH MISSING MAXILLARY PREMOLAR.
Brief Title: Effect Of PRF Versus Xenograft In Closed Sinus Lift.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud adel shaaban (Other)
Responsible Party: Sponsor-Investigator, Mahmoud adel shaaban, CairoU, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo Univ.
Record Dates: First submitted 2018-09-16; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Implant or Graft; Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Patallel Assignment
Who Masked: Investigator
Masking Description: Single investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Used of PRF in clsed sinus lifting (Other): Used of PRF in closed sinus lifting with implant placement
  Interventions: Other: Prf
- Closed sinus with xenograft (No Intervention): used of xenograft in closed sinus lift with implant placement.

INTERVENTIONS:
Other: Prf — Take 10 cc blood from patient and gain prf
  Arms: Used of PRF in clsed sinus lifting

SUMMARY:
Indirect sinus lift with used PRF as a graft material versus xenograft

DETAILED DESCRIPTION:
Crestal incision and reflect the tissue until exposure of the bone, then use drilling to make osteotomy. Then use sutable osteotomes to elevate the sinus floor, then pack of Prf or bone graft in the osteotomy and implant placement . Then closed the flap and suturing.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous area and bone high at least 5-6 mm below the maxillary sinus at maxillary premolar.
* Good oral hygiene.

Exclusion Criteria:

* bad oral hygiene.
* patient with systemic disease that may affect normal healing
* pregnant patients.
* patients with bone diseases and presence of periapical pathology affecting the neighboring teeth.
* Heavy smoker more than 20 cigarettes per day

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Primary stability by ostell device | up to 3 months
  Implant stability will be mesured by ostell device, implant stability will be mesured intra operative at 0 ( time of implant placement ) and 2, 4, 6, 10 and 12 weeks after surgery